CLINICAL TRIAL: NCT02324322
Title: Non-Ambulatory SCI Walk Using a Robotic Exoskeleton: Effect on Bone and Muscle
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kessler Foundation (Other)
Collaborators: New Jersey Commission on Spinal Cord Research (Other)
Responsible Party: Principal Investigator, Gail Forrest, Principal Investigator, Kessler Foundation
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSCR131RG013
Record Dates: First submitted 2014-12-03; First posted 2014-12-24 (Estimated); Last update posted 2017-03-22 (Actual); Status verified 2017-03

CONDITIONS: Spinal Cord Injury
Keywords: Device: Robotic Exoskeleton
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Biopsy, Needle

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Exoskeleton training (Experimental): To examine the effectiveness of robotic exoskeleton-assisted over ground walking (5 hrs. p/wk, 100 sessions, 20 wks = 100 hrs) to induce positive changes in muscle volume and structure of the lower limbs for non-ambulatory persons with SCI. Combined with our current training protocol where people step 1500-2000/session we predict that the 2,000 lower extremity muscle contractions will be sufficient in our proposed exoskeletal study.
  MRI's will be performed to accurately assess muscle CSA of each lower limb to determine individual's muscle thigh and shank volume.
  Muscle Biopsies for the quadricep muscle will be performed to determine changes in BMD and bone structure due to intensive exoskeleton assisted walking.
  Interventions: Device: Exoskeleton Training; Other: Muscle Biopsies; Other: MRI

INTERVENTIONS:
Device: Exoskeleton Training — Exoskeleton Training (100 sessions - 1 hour, 4 - 5 sessions per week for 20 weeks) to enhance functional ambulation for persons with a spinal cord injury. To examine the effectiveness of exoskeleton assisted overground walking to induce positive changes in muscle volume and structure of the lower limbs for non-ambulatory persons with SCI.
  Other Names: Ekso
Other: Muscle Biopsies — Needle Biopsies for Quadricep Muscles will be performed to define changes in BMD and Bone structure with intensive exoskeleton assisted walking. This procedure includes having a trained physician make a small skin incision, after numbing the area over the muscle, and then removing a tiny sliver of muscle to study under the microscope. Three separate biopsies for one incision will be obtained. The biopsies will be performed at baseline, 7 days, and after the intervention.
  To define changes in biochemical markers of bone metabolism with intensive exoskeleton-assisted walking.
  Other Names: Needle Biopsies
Other: MRI — MRI's will provide accurate assessments of muscle CSA of each lower limb (from above the origin of the iliopsoas to the insertion of the achilles tendon) to determine individual's muscle thigh and shank volume.

SUMMARY:
The purpose of this research study is to evaluate an exoskeleton device and mobility skills in the device.

DETAILED DESCRIPTION:
Currently, the treatment of muscle and bone deterioration after SCI is very limited; therefore, there is a definite need to further understand the mechanism of breakdown in the musculoskeletal system after a SCI, and, more importantly, find a clinical strategy that will treat muscle and bone loss.

This pilot research grant will collect results that will be used for the design of a multi-site randomized controlled clinical trial to determine whether a Robotic Exoskeleton training [100 sessions; 1hr/session; 4-5 sessions/week] can improve musculoskeletal outcomes more than other current interventions. If the overall objective is to use the progression of technology to enhance functional ambulation for persons with a spinal cord injury, then the investigators need to evaluate the health benefits associated with continual use of the device.

The study will be a prospective, single-group, repeated measure design using a 2 -month lead in to establish stability, 5-month intervention phase and 2 -month follow-up phase for retention will be performed. Each participant will be used as his or her own control. This project will be completed at two sites: Kessler Foundation will be the lead site that will be under the direction of Dr. Gail F Forrest (Principal Investigator) and Spinal Cord Damage Research Center, James J Peters VA Medical Center under the direction of Dr. Ann M. Spungen (collaborator). Both sites have exoskeletal-assisted walking programs.

ELIGIBILITY:
Inclusion Criteria:

* Must be a non walker with a SCI greater than 1 year post injury
* Must have a neurological level between the C6-T10 level
* Must have a lower extremity score greater than 1 as defined by the neurological exam
* Must be between 21 and 45 years old
* Must be wheelchair reliant 100% of time
* Must have knee bone mineral density greater than .5755 gm/cm2 as determined by study staff
* Must have a score on the Modified Ashworth Scale equal to or less than 3 as determined by the study staff
* Must be able to tolerate upright standing for up to 30 minutes
* Must have joint range of motion within normal functional limits for ambulation
* Must have sufficient upper body strength to balance using the walker while wearing the exoskeleton
* Must have a height between 62 inches or 74 inches
* Must weigh less than 220 lbs,(limitation of the devices)
* Must have no joint tightening of any extremity that limits movement during walking with the assistive devices
* Must have no medical issue that precludes full weight bearing, ambulation or exercise intolerance in the exoskeleton (e.g. orthopedic injuries, pain, severe spasticity)
* Must have no skin issues (e.g. pressure sores) that would prevent wearing the device
* Must have no memory and/or thinking disability (e.g. due to brain injury)
* Must be able to follow directions well and demonstrate learning capability
* Must be able to physically fit into the exoskeletal device

Exclusion Criteria:

* A woman who is pregnant, lactating, or post-menopausal
* Wearing an external device that supports the spinal column or the head, neck, or trunk
* Have persistent orthostatic hypotension (blood pressure drop of more than 30 millimeters of Mercury in robotic system)
* Have had a hospitalization for heart attack, heart surgery or acute heart failure within 3 months of enrollment in study or no presence of major cardiovascular or pulmonary disease, lower extremity deep vein thrombosis (within the last three months)
* Have been taking any medications known to influence bone metabolism

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 13 (Estimated)
Dates: Start 2013-10; Primary Completion 2017-12 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Bilateral Muscle Volume (surrogate for strength)for thigh and shank will be the primary outcome measurement. | 100 hours
  To examine the effectiveness of exoskeleton assisted overground walking (5 hours per week, 100 sessions, 20 weeks = 100 hours) to induce positive changes in muscle volume and structure of the lower limbs for non-ambulatory persons with SCI.

SECONDARY OUTCOMES:
Muscle Activation | 100 hours
  To examine the effect of exoskeletal assisted walking for 100 sessions in increasing further muscle volume through muscle activation to increase muscle size and strength and mitigate the secondary complications that follow SCI.

CONTACTS AND LOCATIONS:
Overall Officials: Gail F Forrest, PhD, Principal Investigator — Kessler Foundation
Locations (1):
- Kessler Foundation, West Orange, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Yes